CLINICAL TRIAL: NCT04798729
Title: COMPARISON OF SENTRIC OCCLUSION DATA OBTAINED FROM TWO DIFFERENT COMPUTER-ASSISTED RECORDING METHODS
Brief Title: Comparison of Two Different Digital Methods in Occlusal Analysis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Evsen Tamam, Assoc Prof Dr, Clinical Professor, Gazi University
Other Study IDs: 2017-419
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Dental Occlusion; Occlusion; Jaw Relationship; Centric Occlusion; Occlusal Analysis
Keywords: Dental Occlusion; Centric Occlusion; Occlusal Analysis; T-Scan; Cerec Omnicam; Digital Dentistry
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Digital Occlusal Recording with T-Scan — Occlusal contact recordings of all the teeth were obtained digitally under conditions of maximum bite force and centric occlusion only with the T-Scan (T-Scan III, version 9.1, Tekscan Inc., South Boston, USA).
Device: Digital Occlusal Recording with Cerec Omnicam — Occlusal contact recordings of all the teeth were obtained digitally under conditions of maximum bite force and centric occlusion only with the CEREC Omnicam™ (version 4.2, Sirona Dental Systems, New York, USA).

SUMMARY:
Aim: The aim of this study is to compare the T-Scan digital occlusal analysis system and the occlusal analysis mode of the CEREC Omnicam system, which is mainly used for design/ production, using the data recorded at the centric occlusion position.

Material-Method: Occlusal recordings were obtained from healthy 20 females and 20 males aged 18-25 at the centric occlusion position. Records were saved as .jpeg format and transferred to Adobe Photoshop CS6 program. Blue, green, and red colors (shown by the same color codes in both systems) representing light, intense and tight contacts, respectively, were evaluated in terms of the pixel counts. For statistical comparison the differences between the systems Independent Sample T-Test and, between the genders, One Sample T- Test were used (α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with no missing teeth (teeth numbers 18, 28, 38, 48 were excluded from the evaluation), no local or systemic disorders that could prevent the bite, and no disorder determined as a result of the TMJ examination.

Exclusion Criteria:

-

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — A total of 20 males and 20 females were included in the study, all aged 18-25 years, with no missing teeth (teeth numbers 18, 28, 38, 48 were excluded from the evaluation), no local or systemic disorders that could prevent the bite, and no disorder determined as a result of the TMJ examination.
Study Population: The groups were formed of voluntary participants from undergraduate and postgraduate students in the Dentistry Faculty of Gazi University.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Comparing the levels of accuracy of the occlusal analysis mode included in the software of CEREC Omnicam and the T-Scan occlusal analysis system. | 6 months
  In both systems, the data of contact intensity were defined with a color scale of blue to red where blue showed the lowest intensity and red the highest. The contact area images obtained from both systems were recorded in .jpeg format and were then transferred to the Adobe Photoshop CS6 program (Adobe Systems, USA) for comparisons to be made.
  The number of pixels in the contact areas of the upper and lower jaws of each subject in all the recordings obtained with the T-Scan and CEREC Omnicam systems were determined using the Adobe Photoshop CS6 pixel-based photographic procedure program.

CONTACTS AND LOCATIONS:
Overall Officials: Evsen TAMAM, Phd, DDS, Assoc Prof Dr, Study Chair — Gazi University Faculty of Dentistry
Locations (1):
- Gazi University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is planned to publish all the collected data as an article in a well-known journal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The study has already been prepared to submit to a journal. It is requested to be published on condition that it is accepted.

REFERENCES:
- [Derived] Bostancioglu SE, Togay A, Tamam E. Comparison of two different digital occlusal analysis methods. Clin Oral Investig. 2022 Feb;26(2):2095-2109. doi: 10.1007/s00784-021-04191-1. Epub 2021 Oct 1. PMID 34596770